CLINICAL TRIAL: NCT07068074
Title: A Randomized Phase III Study of Management of Treatment Naive Primary Melanoma in Elderly Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA6244
Record Dates: First submitted 2025-06-17; First posted 2025-07-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Melanoma
Keywords: A Randomized Phase III Study of Management of Treatment Naive Primary Melanoma in Elderly Patients; cutaneous melanoma; Naive Primary Melanoma in Elderly Patients
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Arm A: WLE and SLN biopsy with surveillance of nodal basin then Surveillance plus Standard of care adjuvant therapy then follow-up Arm B: WLE alone with surveillance of nodal basin then Surveillance plus Standard of care adjuvant therapy then follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): WLE and SLN biopsy with surveillance of nodal basin
  Interventions: Procedure: Sentinel Lymph Node and Wide Local Excision
- Arm B (Experimental): WLE only, with surveillance of nodal basin
  Interventions: Procedure: Wide local Excision

INTERVENTIONS:
Procedure: Wide local Excision — A wide local excision (WLE) is a surgical procedure performed to cut out an abnormal lesion and some surrounding normal tissue.
  Arms: Arm B
Procedure: Sentinel Lymph Node and Wide Local Excision — A wide local excision (WLE) is a surgical procedure performed to cut out an abnormal lesion and some surrounding normal tissue. This is sometimes followed by a sentinel lymph node (SLN) biopsy, in which lymph nodes that cancer cells could spread to are removed as well.
  Arms: Arm A

SUMMARY:
Can we treat your melanoma just as effectively without doing a sentinel lymph node (SLN) biopsy in addition to your wide local excision (WLE) procedure? A wide local excision (WLE) is a surgical procedure performed to cut out an abnormal lesion and some surrounding normal tissue. This is sometimes followed by a sentinel lymph node (SLN) biopsy, in which lymph nodes that cancer cells could spread to are removed as well.

We are doing this study because we want to find out if performing the WLE alone is just as effective as the usual approach for your melanoma, and if it leads to improvements in patients' overall well-being. The usual approach is defined as care most people get for the early stage of melanoma that you currently have.

DETAILED DESCRIPTION:
This study hypothesizes that WLE plus SLN will not significantly change the 2-year recurrence-free survival (RFS) rate compared to WLE alone for elderly patients, and that de-escalated management will result in superior patient-reported outcomes (PRO). The goal of this study is to obtain clinical outcomes data, both RFS and PRO, on older patients who undergo SOC (WLE and SLN biopsy when indicated) vs. de-escalated surgical management [WLE only, without SLN biopsy, with nodal basin surveillance (US or CT, per institutional/physician preference)] of early-stage primary melanoma. A less aggressive treatment approach may spare patients more extensive surgery, more frequent follow up visits, and may result in less frequent utilization of adjuvant therapy, which may be of limited benefit in older/more frail patients with competing causes of mortality. As SLN metastases are less common in the elderly, and this population has competing causes of mortality, we may be over aggressively managing older melanoma patients. The concern becomes that a positive SLN may go undetected in patients randomized to de-escalated care with WLE only, and thus the patient may be under staged (presumed stage I-II when they in fact have occult stage III disease). It is important to note that for patients with clinically occult SLN metastases, 5-year MSS ranges from 93%-32% at 5 years11. In patients who have moderate to severe comorbidities that are likely to interfere with life expectancy within that time frame, or in patients age ≧85, more aggressive measurements may not provide long-term benefit.

Adjuvant immunotherapy with anti-PD1 is approved by the FDA for resected stage IIB/IIC melanoma on the basis of improved RFS13. Thus, patients with stage IIB and higher resected melanoma are now candidates for adjuvant anti-PD1. However, while generally well tolerated, adjuvant immunotherapy is associated with ~15% severe immune related adverse events (IRAEs), for an approximately 50% reduction in recurrence risk. In the clinic, conversations are frequently had with the elderly patient population about whether to pursue SLN and/or adjuvant therapy, though prospective data to address this question are sorely lacking. It is important to note that the goal of this trial is to determine whether SLN biopsy impacts RFS and PRO. This trial does not mandate whether or not physicians utilize adjuvant therapy, which is an option in the current treatment landscape regardless of nodal status (approved for stage IIB-IIID). Data on whether adjuvant therapy is utilized will be captured, and the trial has adequate power to detect differences in RFS and PRO regardless of adjuvant therapy use, as outlined in the statistics section.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 75 years of age.
* Patient must have ECOG Performance Status of 0-2.
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have newly diagnosed primary cutaneous melanoma with wide local excision (WLE) and sentinel lymph node (SLN) biopsy indicated per the treating physician, pending definitive surgical management.
* Patient must be eligible for WLE and SLN biopsy. Patients for whom SLN biopsy would be contraindicated, difficult to perform (i.e., after prior surgery in the draining basin) or impossible (i.e., after prior lymphadenectomy for another cause) are not eligible.
* Patient must be eligible for surgery and not have uncontrolled medical condition that in the opinion of the medical or surgical oncologist precludes surgical management.
* Patient must be English or Spanish speaking to be eligible for this study in order to complete the patient-reported outcomes (PROs). Patients who speak only French can be enrolled in Canada and appropriate documents will be made available by the study team.

Exclusion Criteria:

* Patient must not have an active infection that precludes enrollment to this study in opinion of treating investigator.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome (PRO) Component | (FACT-M) baseline 4 months 8 months 12 months 16 months 20 months 24 months
  The patient reported outcomes (PRO) in this study include a Geriatric Assessment (GA) and the FACT-M Quality of Life (QOL). The National Comprehensive Cancer Network (NCCN) guidelines advocate geriatric assessment (GA) for older patients with cancer to identify health status issues that increase the risk of adverse outcomes. A GA evaluates comorbidity, functional status, physical performance, cognitive ability, psychological status, medications and social support with standardized tools that predict morbidity and mortality in community-dwelling vulnerable older adults. Benefits of GA in community-dwelling vulnerable older adults include prevention of geriatric syndromes, recognition of cognitive deficits, addressing geriatric abnormalities detected by the assessment to prevent hospitalizations and nursing home admissions, and overall improvement of quality of life.

SECONDARY OUTCOMES:
Geriatric Assessment (GA) | Geriatric Assessment (at years 1 and 2 during the surveillance stage and at the time of disease recurrence).
  To evaluate the correlation between geriatric assessment (GA) findings at baseline by domain and study outcomes including RFS, OS, MSS.
  To evaluate the correlation between changes in GA score over the study period and study outcomes including RFS, OS, MSS.
  To use the baseline and follow up GA data to develop an assessment tool to allow for future risk assessment for older adults with early-stage melanoma to guide the decision regarding surgical approach.
  To validate the Geriatric Assessment instrument with data obtained from this study.

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, MD, Study Chair — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States